CLINICAL TRIAL: NCT00664937
Title: A 3 Period, Double-Blind, Randomized Crossover Study to Evaluate the Effects of a Single Dose of Montelukast Compared With Placebo on Exercise-Induced Bronchoconstriction as Assessed by Hyperpolarized Gas Magnetic Resonance Imaging.
Brief Title: Exercise Induced Bronchoconstriction (0476-359)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0476-359; MK0476-359; 2008_502
Record Dates: First submitted 2008-04-22; First posted 2008-04-23 (Estimated); Last update posted 2024-05-09 (Actual); Status verified 2022-01

CONDITIONS: Asthma, Exercise-induced
MeSH Terms: conditions — Asthma, Exercise-Induced | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- I (Placebo Comparator): Three period crossover study, 7 week duration: During periods I-III patients will receive oral medication as a single dose before exercise challenge. For the three periods of this study patients will receive in a randomized sequence one dose of montelukast 10mg and a matching placebo during the other 2 periods.
  Interventions: Drug: montelukast sodium; Drug: Comparator: placebo (unspecified)
- II (Placebo Comparator): Three period crossover study, 7 week duration: During periods I-III patients will receive oral medication as a single dose before exercise challenge. For the three periods of this study patients will receive in a randomized sequence one dose of montelukast 10mg and a matching placebo during the other 2 periods.
  Interventions: Drug: montelukast sodium; Drug: Comparator: placebo (unspecified)
- III (Placebo Comparator): Three period crossover study, 7 week duration: During periods I-III patients will receive oral medication as a single dose before exercise challenge. For the three periods of this study patients will receive in a randomized sequence one dose of montelukast 10mg and a matching placebo during the other 2 periods.
  Interventions: Drug: montelukast sodium; Drug: Comparator: placebo (unspecified)

INTERVENTIONS:
Drug: montelukast sodium — single oral dose, before exercise challenge, of montelukast 10mg; 7 week duration.
  Other Names: MK0476; Singulair®
Drug: Comparator: placebo (unspecified) — single oral dose, before exercise challenge, of Pbo; 7 week duration.

SUMMARY:
Exercise-induced bronchoconstriction (EIB) is a condition where airways tighten when you exercise and may cause coughing, wheezing, or shortness of breath. In many patients, this condition can cause lung function to drop making it harder to breath. An instrument called a spirometer is commonly used to measure lung function. This traditional means of assessing lung function in asthma is limited in its ability to provide information as to where in the lung the tightness is. Hyperpolarized helium magnetic resonance imaging (3He MRI) is a novel way to see the where air is going in the lungs using an MRI and special gas. The ability to see where the air can and cannot reach in the lungs may help show more accurately if a medication is working to make the asthma better. The purpose of this study is to examine patients with EIB in order to see if 3He MRI provides a better way to measure lung function. Patients will be given either montelukast sodium, a drug to improve the ability to breath with EIB, or placebo and then put on a treadmill to induce an occurrence of airway constriction. The patient's lung function will be measured more than once using both the spirometer and the 3He MRI.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a man or woman who is between the ages of 18 and 55 years of age at Visit 1
* Female patients of that are of childbearing potential must show they are not pregnant either by blood test Visit 1 and agree to use appropriate single barrier or hormonal contraception during the course of the study and continuing for at least 14 days following the patient's last study visit
* The patient has stable asthma without any worsening (e.g., requiring unscheduled visit to a physician, hospital or other healthcare resource, new medications or change in dose or frequency of current medications) within 4 weeks of Visit 1 and Visit 2
* Patient is a current non-smoker and if has a history of smoking, has not smoked for at least 6 months and has a smoking history of no more than 15 pack-years (i.e., 1 pack per day for 15 years)

Exclusion Criteria:

* Patient has donated a unit of blood within 4 weeks prior to Visit 1 or anticipates donating blood at any time during this study
* Patient has participated in a clinical trial involving an investigational or marketed medication within the 4 weeks prior to Visit 1 or anticipates participating in any other clinical trial during this study. Patient is currently a regular user, or a recent past abuser (within the past 5 years), of alcohol or illicit drugs
* Patient is a female who has given birth in the last 8 weeks of Visit 1 or breast feeding an infant
* Patient is pregnant, or intends to become pregnant during the time course of the study. Patient is hospitalized or has had a major surgical procedure, major trauma requiring medical attention, or significant illness requiring medical attention within 4 weeks of Visit 1
* Patient does not agree to limit caffeinated beverages and/or chocolate within 8 hours of study visits. Patient has had a worsening of their asthma within 4 weeks of Visit 1 or Visit 2 (i.e., requiring change in type, dose or frequency of medications and/or an unscheduled visit to a health care provider, including emergency room or hospital). Patient has unresolved signs and/or symptoms of an upper respiratory tract infection within 4 weeks of Visit 1 or Visit 2
* Patient is unwilling to restrict vigorous exercise (e.g., weight lifting or long distance running) or abstain from performing strenuous activity within 18 hours of any visit
* Patient has an implanted mechanically, electrically or magnetically activated device or any metal in their body which cannot be removed, including but not limited to: pacemakers, neurostimulators, biostimulators, implanted insulin pumps, aneurysm clips, bioprosthesis, artificial limb, metallic fragment or foreign body, shunt, surgical staples (including clips or metallic sutures) and/or ear implants

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Ventilation volume by 3He MRI, ventilation volume defects by 3He MRI, pulmonary lung function by spirometer | 5 minutes to 1 hour after exercise challenege

SECONDARY OUTCOMES:
Reproducability of ventilation volume and ventilation volume defects as measured by 3He MRI | 3-7 days apart.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: No